CLINICAL TRIAL: NCT00471146
Title: A Randomized, Double-Blind Phase 3 Study Of Gemcitabine Plus AG-013736 Versus Gemcitabine Plus Placebo For The First-Line Treatment Of Patients With Locally Advanced, Unresectable Or Metastatic Pancreatic Cancer.
Brief Title: Study Of Gemcitabine Plus AG-013736 Versus Gemcitabine For Advanced Pancreatic Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4061028
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Randomized Study Of Gemcitabine Plus AG-013736 Versus Gemcitabine Plus Placebo For Advanced Pancreatic Cancer.
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — Axitinib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: AG-013736; Drug: Gemcitabine
- B (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: placebo

INTERVENTIONS:
Drug: AG-013736 — oral administration, starting dose 5 mg twice daily [BID] every day until unacceptable toxicity or tumor progression.
  Arms: A
Drug: Gemcitabine — intravenous administration at 1,000 mg/m^2 day 1, day 8 and day 15 every 4 weeks (conventional dose) until unacceptable toxicity or tumor progression.
  Arms: A
Drug: Gemcitabine — intravenous administration at 1,000 mg/m^2 day 1, day 8 and day 15 every 4 weeks (conventional dose) until unacceptable toxicity or tumor progression.
  Arms: B
Drug: placebo — placebo
  Arms: B

SUMMARY:
The purpose of this study is to determine whether investigational study drug, AG-013736, and gemcitabine are effective in the first-line treatment of advanced pancreatic cancer.

DETAILED DESCRIPTION:
This study was prematurely discontinued for futility on 23 January 2009, based on a planned interim analysis by an independent Data Safety Monitoring Board (DSMB) that found no evidence of improvement in the primary endpoint (survival) in patients treated with axitinib and gemcitabine compared to gemcitabine alone. Enrollment on this study has been discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, metastatic or locally-, advanced pancreatic adenocarcinoma not amenable to curative resection.
* Adequate renal, hepatic and bone marrow function.
* Performance status 0 or 1.

Exclusion Criteria:

* Prior treatment with any systemic chemotherapy for metastatic disease.
* Prior treatment with gemcitabine, AG-013736, or other vascular endothelial growth factor inhibitors.
* Current or recent bleeding, thromboembolic event and or use of a thrombolytic agent.
* Inability to take oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (166):
- United States (60):
  - Pfizer Investigational Site, Antioch, California
  - Pfizer Investigational Site, Corona, California
  - Pfizer Investigational Site, Glendora, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, LaVerne, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Pleasent Hill, California
  - Pfizer Investigational Site, Pomona, California
  - Pfizer Investigational Site, Rancho Cucamonga, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Leandro, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Coeur d'Alene, Idaho
  - Pfizer Investigational Site, Alton, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Beech Grove, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shelbyville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Burlington, Massachusetts
  - Pfizer Investigational Site, Peabody, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Sylvania, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Round Rock, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Lynchburg, Virginia
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Kennewick, Washington
  - Pfizer Investigational Site, Lakewood, Washington
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Argentina (4):
  - Pfizer Investigational Site, Bahía Blanca, Buenos Aires
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Santa Fe, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
- Australia (4):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, East Bentleigh, Victoria
- Austria (3):
  - Pfizer Investigational Site, Salzburg
  - Pfizer Investigational Site, Vienna
  - Pfizer Investigational Site, Wels
- Belgium (4):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Wilrijk
- Canada (9):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- France (8):
  - Pfizer Investigational Site, Clichy
  - Pfizer Investigational Site, La Chaussée-Saint-Victor
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Herblain
- Germany (9):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Greifswald
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Ulm
- Pfizer Investigational Site, Shatin, NT, Hong Kong
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Kaposvár
  - Pfizer Investigational Site, Szentes
  - Pfizer Investigational Site, Zalaegerszeg
- India (5):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Andhra, Pradesh
  - Pfizer Investigational Site, Chennai, Tamil Nadu
- Pfizer Investigational Site, Dublin, Ireland
- Italy (5):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Verona
- Japan (8):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Kashiwa-shi, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Suntougun, Shizuoka
  - Pfizer Investigational Site, Chuo-ku, Tokyo
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam, North Holland
  - Pfizer Investigational Site, Amsterdam
- Russia (5):
  - Pfizer Investigational Site, Moscow, Moscow
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Omsk
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Sochi
- Singapore (2):
  - Pfizer Investigational Site, Singapore, Singapore
  - Pfizer Investigational Site, Singapore
- South Africa (6):
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Observatory
  - Pfizer Investigational Site, Parktown
  - Pfizer Investigational Site, Port Elizabeth
  - Pfizer Investigational Site, Pretoria
  - Pfizer Investigational Site, Sandton
- Pfizer Investigational Site, Seoul, South Korea
- Spain (9):
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Móstoles, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Toledo, Toledo
- Sweden (2):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Uppsala
- Pfizer Investigational Site, Winterthur, Switzerland
- Taiwan (3):
  - Pfizer Investigational Site, Kuei-Shan Jsoamg, Taoyuan County
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- United Kingdom (10):
  - Pfizer Investigational Site, Whitchurch, Cardiff
  - Pfizer Investigational Site, Maidstone, Kent
  - Pfizer Investigational Site, Leicester, Leicestershire
  - Pfizer Investigational Site, Withington, Manchester
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Southhampton

REFERENCES:
- [Derived] Kindler HL, Ioka T, Richel DJ, Bennouna J, Letourneau R, Okusaka T, Funakoshi A, Furuse J, Park YS, Ohkawa S, Springett GM, Wasan HS, Trask PC, Bycott P, Ricart AD, Kim S, Van Cutsem E. Axitinib plus gemcitabine versus placebo plus gemcitabine in patients with advanced pancreatic adenocarcinoma: a double-blind randomised phase 3 study. Lancet Oncol. 2011 Mar;12(3):256-62. doi: 10.1016/S1470-2045(11)70004-3. PMID 21306953
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061028&StudyName=Study%20Of%20Gemcitabine%20Plus%20AG-013736%20Versus%20Gemcitabine%20For%20Advanced%20Pancreatic%20Cancer.

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + Gemcitabine: Axitinib (AG-013736) tablet 5 milligram (mg) orally twice daily (BID) in cycles of 4 weeks. Gemcitabine 1000 mg per square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
- Placebo + Gemcitabine: Placebo matched to axitinib 5 mg tablet orally BID in cycles of 4 weeks. Gemcitabine 1000 mg/m^2 IV infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
Period: Overall Study
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Started | 314 | 316
Treated | 305 | 308
Completed | 142 | 142
Not Completed | 172 | 174
Not completed — Adverse Event | 32 | 33
Not completed — Withdrawal by Subject | 14 | 11
Not completed — Death | 11 | 12
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Objective progression or relapse | 84 | 87
Not completed — Global deterioration of health status | 12 | 14
Not completed — Randomized but not treated | 9 | 8
Not completed — Other | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Axitinib + Gemcitabine: Axitinib (AG-013736) tablet 5 mg orally BID in cycles of 4 weeks. Gemcitabine 1000 mg/m^2 30 minutes IV infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine | Total
Number analyzed (Participants) | 314 | 316 | 630
Age, Customized [Number; unit: Participants]
  Less than 65 years | 203 | 179 | 382
  Greater than or equal to 65 years | 111 | 137 | 248
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 128 | 251
  Male | 191 | 188 | 379

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Time in weeks from randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death or at least 1 year after the randomization of last participant
Population: Intent-to-treat (ITT) population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Weeks | 36.9 [30.1 to 41.1] | 35.8 [30.0 to 44.8]
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Placebo + Gemcitabine; Differences in OS between treatment arms was analyzed by 1-sided log rank test, stratified for extent of disease (locally advanced cancer versus metastatic cancer); Test type: Superiority or Other; p = 0.5436, Log Rank — One-sided log-rank test at alpha = 0.025 significance level was used; Hazard Ratio (HR) = 1.014, 95% CI 2-sided [0.786 to 1.309]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time in weeks from randomization to the first documentation of objective tumor progression or death due to any cause. PFS was calculated as = (first event date minus randomization date plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline until disease progression or at least 1 year after the randomization of last participant
Population: ITT population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Weeks | 19.1 [17.1 to 24.4] | 18.9 [16.2 to 22.6]
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Placebo + Gemcitabine; Differences in PFS between treatment arms was analyzed by 1-sided log rank test, stratified for extent of disease (locally advanced cancer versus metastatic cancer); Test type: Superiority or Other; p = 0.5203, Log Rank — One-sided log-rank test at alpha = 0.025 significance level was used.The p-value was not adjusted for multiple testing; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.779 to 1.298]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: Baseline, every 8 weeks until tumor progression or death
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Percentage of participants | 4.9 [2.5 to 8.3] | 1.6 [0.4 to 4.0]
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Placebo + Gemcitabine; Differences in OR between treatment arms was analyzed by 1-sided Cochran-Mantel-Haenszel (CMH) test, stratified for extent of disease (locally advanced cancer versus metastatic cancer); Test type: Superiority or Other; p = 0.038, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 3.2, 95% CI 2-sided [1.0 to 10.1]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7.
Time Frame: Baseline until death or at least 1 year after the randomization of last participant
Population: DR was calculated for the subgroup of participants from the ITT population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 12 | 4
Weeks | 33.1 [16.1 to 33.1] | NA [NA to NA] — Median duration of response for placebo+gemcitabine arm did not reach at the time of data cut-off.

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Core-30 (EORTC QLQ- C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status (GHS), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0- 100 scale; higher score=better level of functioning or greater degree of symptoms. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Baseline, Day 1 (D1) of each cycle (C2-C13) up to 28 days after the last dose (follow-up) or early withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Units on a scale
  Physical functioning: Baseline (n=295, 289) | 77.445 (20.3052) | 78.546 (18.9192)
  Physical functioning: Change at C2 D1 (n=233, 233) | -2.713 (16.7682) | -3.261 (15.0742)
  Physical functioning: Change at C3 D1 (n=173, 179) | -5.897 (19.3522) | -1.565 (16.2738)
  Physical functioning: Change at C4 D1 (n=134, 133) | -5.671 (18.8623) | -1.453 (17.1209)
  Physical functioning: Change at C5 D1 (n=96, 82) | -2.498 (21.8687) | -0.076 (16.9709)
  Physical functioning: Change at C6 D1 (n=59, 58) | -5.193 (19.6995) | -1.719 (15.5260)
  Physical functioning: Change at C7 D1 (n=38, 37) | -1.924 (14.2726) | 0.011 (18.9261)
  Physical functioning: Change at C8 D1 (n=15, 21) | -4.000 (16.8759) | 0.014 (13.8428)
  Physical functioning: Change at C9 D1 (n=9, 9) | 0.033 (15.2534) | -12.578 (20.9490)
  Physical functioning: Change at C10 D1 (n=3, 4) | 6.667 (17.5754) | -1.675 (22.0563)
  Physical functioning: Change at C11 D1 (n=1, 1) | 0.000 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -6.600 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Physical functioning: Change at C12 D1 (n=1, 0) | 0.000 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Physical functioning: Change at C13 D1 (n=1, 0) | 0.000 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Physical functioning:Change at followup (n=67, 70) | -17.713 (23.8263) | -11.523 (21.0513)
  Role functioning: Baseline (n=297, 295) | 66.3 (30.09) | 68.1 (30.72)
  Role functioning: Change at C2 D1 (n=239, 242) | -2.2 (30.95) | -2.8 (25.75)
  Role functioning: Change at C3 D1 (n=177, 185) | -4.6 (32.65) | 1.5 (26.90)
  Role functioning: Change at C4 D1 (n=135, 136) | -4.3 (32.13) | 1.2 (27.18)
  Role functioning: Change at C5 D1 (n=99, 81) | -0.5 (34.95) | -2.7 (29.63)
  Role functioning: Change at C6 D1 (n=60, 58) | -4.4 (29.25) | -2.3 (24.27)
  Role functioning: Change at C7 D1 (n=38, 37) | -3.1 (25.07) | -1.3 (26.75)
  Role functioning: Change at C8 D1 (n=16, 21) | -6.2 (20.05) | 0.0 (31.63)
  Role functioning: Change at C9 D1 (n=9, 9) | 1.9 (28.21) | -20.4 (33.11)
  Role functioning: Change at C10 D1 (n=3, 4) | 5.6 (9.64) | -4.2 (28.46)
  Role functioning: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -50.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Role functioning: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Role functioning: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Role functioning: Change at follow-up (n=66, 72) | -20.0 (31.52) | -14.1 (32.34)
  Emotional functioning (EF): Baseline (n=294, 287) | 70.8 (22.01) | 71.7 (22.47)
  EF: Change at C2 D1 (n=233, 229) | 5.0 (21.48) | 5.0 (18.92)
  EF: Change at C3 D1 (n=170, 180) | 3.7 (20.19) | 3.4 (18.95)
  EF: Change at C4 D1 (n=134, 131) | 3.0 (22.54) | 5.2 (21.12)
  EF: Change at C5 D1 (n=96, 80) | 4.3 (21.09) | 5.9 (17.24)
  EF: Change at C6 D1 (n=60, 56) | 4.0 (19.31) | 6.7 (17.43)
  EF: Change at C7 D1 (n=37, 34) | 0.0 (18.84) | 3.2 (16.28)
  EF: Change at C8 D1 (n=17, 19) | -2.9 (22.05) | 5.3 (14.74)
  EF: Change at C9 D1 (n=9, 9) | 3.7 (16.72) | -4.6 (15.07)
  EF: Change at C10 D1 (n=3, 4) | 13.9 (12.73) | 2.1 (18.50)
  EF: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -16.6 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EF: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  EF: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  EF: Change at follow-up (n=65, 71) | -7.3 (23.51) | -2.7 (23.14)
  Cognitive Functioning (CF): Baseline (n=293, 288) | 78.7 (22.26) | 80.9 (21.50)
  CF: Change at C2 D1 (n=234, 234) | -1.1 (19.86) | -0.3 (17.74)
  CF: Change at C3 D1 (n=172, 179) | -2.1 (20.43) | -0.9 (18.67)
  CF: Change at C4 D1 (n=134, 134) | -4.2 (19.98) | 2.0 (18.62)
  CF: Change at C5 D1 (n=97, 80) | -1.4 (20.21) | 1.7 (18.86)
  CF: Change at C6 D1 (n=60, 56) | -3.1 (19.27) | -4.5 (19.97)
  CF: Change at C7 D1 (n=38, 34) | -4.4 (18.45) | 0.5 (14.50)
  CF: Change at C8 D1 (n=17, 17) | -8.8 (22.15) | -2.9 (23.74)
  CF: Change at C9 D1 (n=9, 9) | -0.0 (25.03) | -1.8 (24.22)
  CF: Change at C10 D1 (n=3, 4) | -5.6 (9.64) | 8.3 (28.88)
  CF: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CF: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  CF: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  CF: Change at follow-up (n=65, 71) | -12.6 (25.01) | -7.5 (25.47)
  Social functioning: Baseline (n=289, 286) | 68.9 (27.98) | 69.7 (28.83)
  Social functioning: Change at C2 D1 (n=232, 230) | 1.3 (24.73) | 0.9 (26.35)
  Social functioning: Change at C3 D1 (n=169, 178) | -1.3 (29.38) | 3.2 (27.31)
  Social functioning: Change at C4 D1 (n=132, 134) | 0.1 (25.51) | 0.6 (26.83)
  Social functioning: Change at C5 D1 (n=95, 80) | 2.1 (27.31) | 0.8 (27.93)
  Social functioning: Change at C6 D1 (n=58, 56) | -4.9 (28.79) | 1.5 (29.52)
  Social functioning: Change at C7 D1 (n=37, 35) | -5.4 (20.05) | 2.4 (29.47)
  Social functioning: Change at C8 D1 (n=17, 19) | 4.9 (29.91) | -1.7 (27.72)
  Social functioning: Change at C9 D1 (n=9, 9) | -0.0 (32.29) | -1.8 (28.20)
  Social functioning: Change at C10 D1 (n=3, 4) | 5.6 (9.64) | 12.5 (43.83)
  Social functioning: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 33.4 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Social functioning: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Social functioning: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Social functioning: Change at follow-up (n=64, 70) | -13.3 (33.75) | -2.6 (33.88)
  Fatigue: Baseline (n=293, 289) | 41.0 (23.87) | 40.1 (25.12)
  Fatigue: Change at C2 D1 (n=227, 228) | 2.8 (21.15) | 2.1 (20.12)
  Fatigue: Change at C3 D1 (n=170, 181) | 3.4 (21.94) | -0.9 (21.76)
  Fatigue: Change at C4 D1 (n=132, 132) | 5.6 (23.97) | -1.1 (22.77)
  Fatigue: Change at C5 D1 (n=97, 80) | -0.0 (24.39) | 1.1 (21.92)
  Fatigue: Change at C6 D1 (n=60, 57) | 5.0 (21.31) | 0.0 (21.22)
  Fatigue: Change at C7 D1 (n=38, 36) | 1.8 (20.61) | 2.2 (19.12)
  Fatigue: Change at C8 D1 (n=17, 20) | 7.2 (22.89) | 4.4 (22.05)
  Fatigue: Change at C9 D1 (n=9, 9) | -6.2 (21.63) | 14.8 (24.21)
  Fatigue: Change at C10 D1 (n=3, 4) | -11.1 (19.28) | -5.5 (27.98)
  Fatigue: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 11.1 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Fatigue: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Fatigue: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Fatigue: Change at follow-up (n=63, 71) | 13.1 (25.93) | 12.1 (25.95)
  Nausea and vomiting: Baseline (n=295, 294) | 12.9 (19.19) | 13.1 (19.75)
  Nausea and vomiting: Change at C2 D1 (n=238, 239) | 3.7 (20.69) | 2.9 (22.93)
  Nausea and vomiting: Change at C3 D1 (n=176, 185) | 1.9 (20.38) | -0.4 (19.54)
  Nausea and vomiting: Change at C4 D1 (n=133, 135) | 3.5 (20.82) | 0.4 (19.68)
  Nausea and vomiting: Change at C5 D1 (n=98, 81) | 4.6 (22.16) | 1.0 (18.88)
  Nausea and vomiting: Change at C6 D1 (n=60, 59) | 6.9 (22.61) | 2.8 (20.33)
  Nausea and vomiting: Change at C7 D1 (n=38, 37) | 1.3 (19.52) | 2.7 (20.24)
  Nausea and vomiting: Change at C8 D1 (n=17, 21) | -4.9 (18.41) | 0.8 (22.66)
  Nausea and vomiting: Change at C9 D1 (n=9, 9) | -13.0 (32.02) | -5.6 (18.64)
  Nausea and vomiting: Change at C10 D1 (n=3, 4) | -11.1 (19.23) | 8.3 (9.58)
  Nausea and vomiting: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Nausea and vomiting: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Nausea and vomiting: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Nausea and vomiting: Change at followup (n=68, 73) | 9.8 (25.63) | 7.5 (22.40)
  Pain: Baseline (n=291, 291) | 40.7 (30.16) | 36.9 (29.57)
  Pain: Change at C2 D1 (n=231, 234) | -10.1 (29.47) | -7.9 (25.28)
  Pain: Change at C3 D1 (n=169, 181) | -13.6 (29.81) | -11.2 (26.63)
  Pain: Change at C4 D1 (n=131, 135) | -12.2 (32.48) | -7.8 (27.14)
  Pain: Change at C5 D1 (n=97, 80) | -10.5 (32.75) | -6.9 (26.21)
  Pain: Change at C6 D1 (n=59, 58) | -11.9 (27.51) | -7.5 (29.48)
  Pain: Change at C7 D1 (n=38, 35) | -14.0 (27.81) | -9.5 (24.67)
  Pain: Change at C8 D1 (n=17, 20) | -9.8 (26.39) | -6.7 (29.32)
  Pain: Change at C9 D1 (n=9, 9) | -22.2 (43.29) | -5.6 (39.08)
  Pain: Change at C10 D1 (n=3, 4) | -33.3 (33.30) | -4.2 (45.88)
  Pain: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pain: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pain: Change at follow-up (n=66, 72) | 3.3 (37.01) | 3.5 (31.14)
  Dyspnoea: Baseline (n=295, 295) | 16.1 (22.30) | 14.8 (23.55)
  Dyspnoea: Change at C2 D1 (n=238, 240) | 5.5 (23.58) | 2.1 (20.91)
  Dyspnoea: Change at C3 D1 (n=175, 186) | 5.7 (26.84) | 3.9 (24.67)
  Dyspnoea: Change at C4 D1 (n=135, 135) | 7.7 (26.99) | 4.4 (21.08)
  Dyspnoea: Change at C5 D1 (n=98, 82) | 4.4 (26.05) | 2.8 (18.29)
  Dyspnoea: Change at C6 D1 (n=60, 59) | 9.4 (26.09) | -0.0 (16.37)
  Dyspnoea: Change at C7 D1 (n=37, 37) | 6.3 (24.63) | 5.4 (20.05)
  Dyspnoea: Change at C8 D1 (n=16, 21) | 4.2 (20.62) | 12.7 (24.66)
  Dyspnoea: Change at C9 D1 (n=9, 9) | 11.1 (47.14) | 14.8 (29.39)
  Dyspnoea: Change at C10 D1 (n=3, 4) | -11.1 (50.92) | 0.0 (27.19)
  Dyspnoea: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Dyspnoea: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Dyspnoea: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Dyspnoea: Change at follow-up (n=68, 73) | 13.2 (28.30) | 8.7 (24.23)
  Insomnia: Baseline (n=297, 295) | 36.8 (31.95) | 32.2 (32.17)
  Insomnia: Change at C2 D1 (n=240, 241) | -13.6 (33.55) | -7.3 (33.16)
  Insomnia: Change at C3 D1 (n=178, 185) | -13.5 (33.33) | -8.7 (33.30)
  Insomnia: Change at C4 D1 (n=134, 134) | -12.7 (38.52) | -11.2 (27.41)
  Insomnia: Change at C5 D1 (n=99, 82) | -14.5 (33.05) | -7.3 (28.70)
  Insomnia: Change at C6 D1 (n=60, 59) | -8.3 (30.46) | -2.3 (30.86)
  Insomnia: Change at C7 D1 (n=37, 37) | -11.7 (36.19) | -2.7 (19.84)
  Insomnia: Change at C8 D1 (n=17, 21) | 5.9 (35.82) | -3.2 (20.82)
  Insomnia: Change at C9 D1 (n=9, 9) | -14.8 (24.23) | -0.0 (23.56)
  Insomnia: Change at C10 D1 (n=3, 4) | 11.1 (19.23) | -0.0 (27.23)
  Insomnia: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Insomnia: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Insomnia: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Insomnia: Change at follow-up (n=68, 73) | 1.5 (36.63) | 1.4 (28.02)
  Loss of appetite: Baseline (n=297, 295) | 39.6 (35.49) | 37.5 (33.36)
  Loss of appetite: Change at C2 D1 (n=240, 240) | -2.1 (34.24) | -2.6 (27.91)
  Loss of appetite: Change at C3 D1 (n=178, 186) | -1.3 (31.57) | -5.9 (31.50)
  Loss of appetite: Change at C4 D1 (n=135, 135) | 0.0 (35.27) | -6.7 (29.88)
  Loss of appetite: Change at C5 D1 (n=99, 82) | 1.7 (35.76) | -4.5 (30.44)
  Loss of appetite: Change at C6 D1 (n=60, 59) | 2.8 (33.22) | -4.5 (29.34)
  Loss of appetite: Change at C7 D1 (n=38, 37) | 0.9 (35.92) | -7.2 (27.37)
  Loss of appetite: Change at C8 D1 (n=17, 20) | 7.8 (25.07) | -1.7 (29.57)
  Loss of appetite: Change at C9 D1 (n=9, 9) | -14.8 (29.41) | -7.4 (36.44)
  Loss of appetite: Change at C10 D1 (n=3, 4) | -22.2 (19.23) | 0.0 (38.48)
  Loss of appetite: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Loss of appetite: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Loss of appetite: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Loss of appetite: Change at follow-up (n=67, 73) | 7.0 (39.17) | 7.8 (36.24)
  Constipation: Baseline (n=293, 289) | 30.7 (32.13) | 29.6 (32.66)
  Constipation: Change at C2 D1 (n=234, 235) | -4.8 (32.18) | -2.8 (33.21)
  Constipation: Change at C3 D1 (n =173, 181) | -7.3 (32.12) | -6.1 (36.43)
  Constipation: Change at C4 D1 (n=134, 135) | -6.5 (35.99) | -10.6 (36.80)
  Constipation: Change at C5 D1 (n=97, 80) | -11.0 (33.59) | -8.7 (29.88)
  Constipation: Change at C6 D1 (n=60, 58) | -5.6 (37.42) | -9.8 (32.45)
  Constipation: Change at C7 D1 (n=38, 36) | -2.6 (31.37) | -13.0 (32.15)
  Constipation: Change at C8 D1 (n=17, 20) | 0.0 (28.87) | -16.7 (39.74)
  Constipation: Change at C9 D1 (n=9, 9) | -18.5 (33.79) | -29.6 (35.14)
  Constipation: Change at C10 D1 (n=3, 4) | -11.1 (19.23) | -50.0 (43.04)
  Constipation: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Constipation: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Constipation: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Constipation: Change at follow-up (n=66, 71) | 5.1 (42.27) | -6.1 (35.77)
  Diarrhoea: Baseline (n=294, 290) | 14.3 (21.68) | 13.7 (24.19)
  Diarrhoea: Change at C2 D1 (n=235, 235) | 1.7 (25.73) | 0.3 (21.78)
  Diarrhoea: Change at C3 D1 (n=173, 182) | 9.4 (28.66) | 0.2 (23.10)
  Diarrhoea: Change at C4 D1 (n=134, 136) | 7.7 (28.00) | -1.5 (22.53)
  Diarrhoea: Change at C5 D1 (n=96, 81) | 11.8 (27.35) | 1.2 (27.10)
  Diarrhoea: Change at C6 D1 (n=60, 58) | 20.0 (33.72) | 1.7 (28.22)
  Diarrhoea: Change at C7 D1 (n=38, 36) | 14.9 (32.60) | 2.8 (23.05)
  Diarrhoea: Change at C8 D1 (n=17, 20) | 25.5 (38.24) | 1.7 (27.52)
  Diarrhoea: Change at C9 D1 (n=9, 9) | 37.0 (45.47) | 22.2 (33.35)
  Diarrhoea: Change at C10 D1 (n=3, 4) | 22.2 (50.91) | 16.7 (19.23)
  Diarrhoea: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Diarrhoea: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Diarrhoea: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Diarrhoea: Change at follow-up (n=66, 71) | 2.5 (29.41) | 2.8 (25.03)
  Financial difficulties (FD): Baseline (n=292, 285) | 24.7 (30.41) | 23.0 (30.83)
  FD:Change at C2 D1 (n=233, 228) | -3.1 (22.95) | -4.5 (23.29)
  FD: Change at C3 D1 (n=171, 176) | -7.2 (26.94) | -3.4 (23.39)
  FD: Change at C4 D1 (n=133, 133) | -5.5 (26.33) | -3.3 (23.52)
  FD: Change at C5 D1 (n=96, 80) | -4.9 (21.62) | 1.3 (25.68)
  FD: Change at C6 D1 (n=60, 56) | -3.9 (24.61) | -1.8 (28.02)
  FD: Change at C7 D1 (n=37, 34) | -2.7 (24.06) | -3.9 (32.60)
  FD: Change at C8 D1 (n=17, 17) | 2.0 (14.28) | 2.0 (34.31)
  FD: Change at C9 D1 (n=9, 9) | 7.4 (22.23) | 3.7 (45.49)
  FD: Change at C10 D1 (n=3, 4) | 0.0 (0.00) | 25.0 (41.94)
  FD: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FD: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  FD: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  FD: Change at follow-up (n=65, 70) | 6.7 (29.59) | -0.5 (21.61)
  GHS/Quality of Life (QoL): Baseline (n=292, 288) | 54.2 (22.34) | 57.1 (23.14)
  GHS/QoL:Change at C2 D1 (n=234, 233) | 2.2 (23.36) | 1.9 (22.39)
  GHS/QoL:Change at C3 D1 (n=168, 180) | -0.3 (25.42) | 5.7 (21.45)
  GHS/QoL:Change at C4 D1(n=132, 132) | 0.1 (23.79) | 2.8 (21.54)
  GHS/QoL:Change at C5 D1 (n=96, 81) | 1.5 (22.63) | 2.7 (18.35)
  GHS/QoL:Change at C6 D1 (n=60, 57) | 0.8 (21.41) | 3.2 (23.40)
  GHS/QoL:Change at C7 D1 (n=38, 35) | 2.6 (23.01) | 2.1 (22.35)
  GHS/QoL:Change at C8 D1 (n=17, 19) | -1.0 (23.73) | 1.3 (23.76)
  GHS/QoL:Change at C9 D1 (n=9, 9) | 7.4 (16.89) | -8.3 (20.39)
  GHS/QoL: Change at C10 D1 (n=3, 4) | 22.3 (19.28) | -0.0 (32.59)
  GHS/QoL: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  GHS/QoL: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  GHS/QoL: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  GHS/QoL:Change at follow-up (n=65, 71) | -9.1 (26.06) | -6.7 (24.50)

6. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Pancreatic 26 (EORTC QLQ- PAN26) Score
Description: QLQ-PAN26 consists of 26 questions (Qs) relating to disease symptoms, treatment (Tx) side effects and emotional issues specific to pancreatic cancer (PC). Questions include on altered bowel habits, pain, dietary changes, disease and Tx-related symptoms and issues related to the emotional and social well-being of participants with PC. All 26 Qs are answered on 4-point Likert scale ranging from '1=not at all' to 4='very much' and subsequently transformed into scales that range from 0-100; higher scores= greater degree of symptoms or treatment side effects and emotional issues.
Time Frame: Baseline, Day 1 (D1) of each cycle (C2-C13) up to 28 days after the last dose (follow-up) or early withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Units on a scale
  Pancreatic Pain: Baseline (n=246, 250) | 41.6 (27.16) | 40.0 (25.54)
  Pancreatic Pain: Change at C2 D1 (n=191, 197) | -10.9 (24.38) | -10.1 (22.93)
  Pancreatic Pain: Change at C3 D1 (n=141, 153) | -16.3 (25.51) | -11.2 (24.92)
  Pancreatic Pain: Change at C4 D1 (n=99, 111) | -13.2 (28.70) | -11.4 (26.16)
  Pancreatic Pain: Change at C5 D1 (n=67, 64) | -15.8 (28.06) | -13.0 (23.85)
  Pancreatic Pain: Change at C6 D1 (n=41, 43) | -15.9 (25.47) | -13.0 (24.62)
  Pancreatic Pain: Change at C7 D1 (n=25, 25) | -15.3 (28.02) | -15.0 (25.69)
  Pancreatic Pain: Change at C8 D1 (n=11, 11) | -7.6 (27.76) | -9.8 (30.01)
  Pancreatic Pain: Change at C9 D1 (n=6, 6) | -29.2 (31.06) | 0.0 (15.81)
  Pancreatic Pain: Change at C10 D1 (n=2, 3) | -20.9 (29.49) | 5.6 (26.79)
  Pancreatic Pain: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pancreatic Pain: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pancreatic Pain: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pancreatic Pain: Change at follow-up (n=47, 46) | -3.5 (29.59) | -3.6 (28.80)
  Hepatic: Baseline (n=245, 254) | 10.2 (17.21) | 10.8 (17.59)
  Hepatic: Change at C2 D1 (n=193, 205) | 0.3 (18.24) | -2.0 (17.67)
  Hepatic: Change at C3 D1 (n=142, 157) | -1.4 (16.78) | -2.5 (18.60)
  Hepatic: Change at C4 D1 (n=99, 112) | -2.5 (18.34) | -2.4 (18.15)
  Hepatic: Change at C5 D1 (n=68, 64) | 1.0 (17.49) | -2.6 (16.60)
  Hepatic: Change at C6 D1 (n=40, 41) | 0.4 (15.34) | -3.2 (17.57)
  Hepatic: Change at C7 D1 (n=25, 24) | -0.7 (16.30) | -4.9 (18.70)
  Hepatic: Change at C8 D1 (n=11, 12) | -4.5 (13.10) | -4.2 (12.57)
  Hepatic: Change at C9 D1 (n=6, 5) | -11.1 (13.60) | -13.3 (13.94)
  Hepatic: Change at C10 D1 (n=2, 2) | -16.7 (23.55) | -8.4 (11.81)
  Hepatic: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Hepatic: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Hepatic: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Hepatic: Change at follow-up (n=47, 48) | 2.8 (23.38) | -1.4 (23.27)
  Digestive Symptom: Baseline (n=250, 255) | 34.3 (30.78) | 33.9 (31.05)
  Digestive Symptom: Change at C2 D1 (n=195, 206) | 2.8 (29.15) | 0.6 (26.72)
  Digestive Symptom: Change at C3 D1 (n=144, 159) | -1.2 (31.58) | -4.3 (32.97)
  Digestive Symptom: Change at C4 D1 (n=100, 114) | 0.5 (30.57) | -4.5 (30.90)
  Digestive Symptom: Change at C5 D1 (n=69, 65) | 1.4 (32.80) | -3.6 (36.14)
  Digestive Symptom: Change at C6 D1 (n=40, 45) | 3.3 (30.23) | 0.4 (35.97)
  Digestive Symptom: Change at C7 D1 (n=25, 26) | -6.0 (30.76) | -1.3 (24.91)
  Digestive Symptom: Change at C8 D1 (n=11, 14) | 4.5 (42.87) | 17.9 (23.07)
  Digestive Symptom: Change at C9 D1 (n=6, 6) | -13.9 (46.44) | 22.2 (25.10)
  Digestive Symptom: Change at C10 D1 (n=2, 3) | -33.3 (47.09) | 11.1 (19.23)
  Digestive Symptom: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Digestive Symptom: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Digestive Symptom: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Digestive Symptom: Change at follow-up (n=47, 47) | 6.0 (38.14) | 2.8 (35.83)
  Sexuality: Baseline (n=217, 232) | 56.8 (36.90) | 55.5 (38.04)
  Sexuality: Change at C2 D1 (n=157, 181) | -0.5 (37.81) | -4.0 (33.17)
  Sexuality: Change at C3 D1 (n=118, 139) | -4.9 (37.70) | -3.0 (32.25)
  Sexuality: Change at C4 D1 (n=85, 100) | -4.1 (38.40) | 3.0 (29.90)
  Sexuality: Change at C5 D1 (n=55, 58) | -1.5 (34.30) | -5.2 (29.32)
  Sexuality: Change at C6 D1 (n=30, 38) | 12.2 (29.67) | -11.4 (33.58)
  Sexuality: Change at C7 D1 (n=19, 21) | 4.4 (35.06) | -7.1 (31.88)
  Sexuality: Change at C8 D1 (n=8, 10) | 12.5 (24.82) | -15.0 (26.59)
  Sexuality: Change at C9 D1 (n=4, 6) | 25.0 (31.93) | 0.0 (23.55)
  Sexuality: Change at C10 D1 (n=0, 3) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | 11.1 (19.28)
  Sexuality: Change at C11 D1 (n=0, 1) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Sexuality: Change at C12 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Sexuality: Change at C13 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Sexuality: Change at follow-up (n=36, 41) | -3.2 (41.18) | -23.2 (42.31)
  Health care(HC)satisfaction: Baseline (n=241, 247) | 78.0 (26.66) | 78.3 (23.94)
  HC satisfaction: Change at C2 D1 (n=182, 194) | 0.1 (27.73) | 1.8 (24.13)
  HC satisfaction: Change at C3 D1 (n=135, 149) | 0.2 (31.54) | 5.4 (24.98)
  HC satisfaction: Change at C4 D1 (n=97, 108) | -4.3 (34.88) | -0.2 (26.52)
  HC satisfaction: Change at C5 D1 (n=66, 59) | 1.0 (29.66) | 0.8 (28.77)
  HC satisfaction: Change at C6 D1 (n=40, 39) | -6.7 (26.91) | -0.4 (27.96)
  HC satisfaction: Change at C7 D1 (n=27, 20) | -4.3 (22.44) | 6.7 (33.06)
  HC satisfaction: Change at C8 D1 (n=12, 11) | -16.7 (52.23) | 7.6 (20.22)
  HC satisfaction: Change at C9 D1 (n=6, 6) | 16.7 (47.14) | -5.6 (17.23)
  HC satisfaction: Change at C10 D1 (n=2, 3) | -33.3 (0.0) | 5.6 (9.64)
  HC satisfaction: Change at C11 D1 (n=1, 1) | -33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  HC satisfaction: Change at C12 D1 (n=1, 0) | -33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  HC satisfaction: Change at C13 D1(n=1, 0) | -33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  HC satisfaction: Change at follow-up (n=46, 45) | -0.7 (29.39) | -2.2 (31.50)
  Body Image: Baseline (n=249, 251) | 28.5 (28.46) | 28.8 (28.67)
  Body Image: Change at C2 D1 (n=189, 200) | 4.9 (23.11) | -0.2 (26.78)
  Body Image: Change at C3 D1 (n=142, 149) | 4.9 (22.26) | 2.1 (26.16)
  Body Image: Change at C4 D1 (n=97, 111) | 6.7 (26.20) | 0.9 (26.48)
  Body Image: Change at C5 D1 (n=70, 62) | 4.8 (26.33) | -0.3 (25.87)
  Body Image: Change at C6 D1 (n=40, 42) | 8.3 (28.24) | -0.8 (33.92)
  Body Image: Change at C7 D1 (n=25, 24) | 12.0 (27.43) | -5.6 (33.22)
  Body Image: Change at C8 D1 (n=11, 12) | 21.2 (42.23) | 11.1 (32.04)
  Body Image: Change at C9 D1 (n=6, 6) | 33.3 (52.69) | 8.3 (46.87)
  Body Image: Change at C10 D1 (n=2, 3) | -8.3 (11.74) | 5.6 (78.77)
  Body Image: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -50.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Body Image: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Body Image: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Body Image: Change at follow-up (n=47, 45) | 13.1 (30.67) | 11.5 (24.56)
  Altered Bowel Habit: Baseline (n=250, 255) | 20.3 (22.92) | 21.2 (25.72)
  Altered Bowel Habit: Change at C2 D1 (n=193, 204) | 3.0 (24.19) | 1.5 (22.21)
  Altered Bowel Habit: Change at C3 D1 (n=143, 156) | 6.2 (26.37) | 2.5 (24.67)
  Altered Bowel Habit: Change at C4 D1 (n=98, 114) | 6.6 (25.52) | 4.8 (22.14)
  Altered Bowel Habit: Change at C5 D1 (n=68, 63) | 8.3 (33.15) | 1.3 (24.56)
  Altered Bowel Habit: Change at C6 D1 (n=40, 43) | 9.6 (30.63) | 2.3 (28.07)
  Altered Bowel Habit: Change at C7 D1 (n=25, 25) | 6.0 (25.40) | 1.3 (30.77)
  Altered Bowel Habit: Change at C8 D1 (n=11, 13) | 1.5 (29.29) | 7.7 (38.86)
  Altered Bowel Habit: Change at C9 D1 (n=6, 6) | 13.9 (32.35) | -5.6 (51.27)
  Altered Bowel Habit: Change at C10 D1 (n=2, 3) | -8.3 (35.36) | -16.7 (72.62)
  Altered Bowel Habit: Change at C11 D1 (n=1, 1) | 16.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -100.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Altered Bowel Habit: Change at C12 D1 (n=1, 0) | 16.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Altered Bowel Habit: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Altered Bowel Habit: Change at followup (n=47, 48) | 6.0 (29.36) | 5.9 (21.33)
  Ascites: Baseline (n=250, 256) | 38.7 (32.98) | 32.9 (30.61)
  Ascites: Change at C2 D1 (n=197, 207) | -8.6 (33.32) | -3.4 (29.65)
  Ascites: Change at C3 D1 (n=144, 158) | -8.3 (33.34) | -5.1 (28.70)
  Ascites: Change at C4 D1 (n=101, 114) | -5.0 (36.64) | -0.3 (26.05)
  Ascites: Change at C5 D1 (n=71, 65) | -8.5 (34.15) | -0.5 (29.17)
  Ascites: Change at C6 D1 (n=42, 45) | -3.2 (31.08) | -2.2 (32.10)
  Ascites: Change at C7 D1 (n=26, 26) | -14.1 (32.91) | -12.8 (23.25)
  Ascites: Change at C8 D1 (n=11, 14) | -18.2 (43.12) | -11.9 (28.05)
  Ascites: Change at C9 D1 (n=6, 6) | -11.1 (34.42) | -16.7 (34.95)
  Ascites: Change at C10 D1 (n=2, 3) | -16.7 (23.55) | 22.2 (38.51)
  Ascites: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Ascites: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Ascites: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Ascites: Change at follow-up (n=48, 48) | 5.6 (35.96) | -2.1 (26.11)
  Indigestion: Baseline (n=252, 257) | 29.4 (30.38) | 24.0 (28.55)
  Indigestion: Change at C2 D1 (n=198, 208) | -0.3 (26.87) | -2.4 (24.29)
  Indigestion: Change at C3 D1 (n=144, 159) | 0.2 (30.16) | -5.2 (25.59)
  Indigestion: Change at C4 D1 (n=101, 115) | -4.0 (24.63) | -4.1 (25.80)
  Indigestion: Change at C5 D1 (n=71, 65) | 0.5 (29.01) | -4.6 (22.72)
  Indigestion: Change at C6 D1 (n=41, 45) | 1.6 (31.58) | -1.5 (24.57)
  Indigestion: Change at C7 D1 (n=26, 26) | -3.8 (19.60) | -1.3 (17.59)
  Indigestion: Change at C8 D1 (n=11, 14) | 0.0 (21.06) | 2.4 (20.53)
  Indigestion: Change at C9 D1 (n=6, 6) | -5.6 (25.07) | 11.1 (27.23)
  Indigestion: Change at C10 D1 (n=2, 3) | -16.7 (23.55) | 22.2 (19.23)
  Indigestion: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Indigestion: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Indigestion: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Indigestion: Change at follow-up (n=48, 48) | 7.6 (30.94) | 1.4 (30.73)
  Flatulence: Baseline (n=249, 256) | 37.9 (32.34) | 34.0 (31.31)
  Flatulence: Change at C2 D1 (n=197, 206) | 1.2 (29.81) | 2.6 (31.82)
  Flatulence: Change at C3 D1 (n=146, 159) | 3.2 (33.07) | 0.2 (34.48)
  Flatulence: Change at C4 D1 (n=101, 115) | -1.3 (33.65) | 2.3 (32.07)
  Flatulence: Change at C5 D1 (n=70, 65) | -1.0 (32.60) | 1.0 (31.17)
  Flatulence: Change at C6 D1 (n=41, 45) | -1.6 (26.83) | -1.5 (29.27)
  Flatulence: Change at C7 D1 (n=25, 26) | -1.3 (26.31) | -3.8 (23.71)
  Flatulence: Change at C8 D1 (n=10, 14) | -10.0 (35.34) | 2.4 (27.62)
  Flatulence: Change at C9 D1 (n=5, 6) | 0.0 (0.00) | 5.6 (13.59)
  Flatulence: Change at C10 D1 (n=1, 3) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -11.1 (19.23)
  Flatulence: Change at C11 D1 (n=0, 1) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Flatulence: Change at C12 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Flatulence: Change at C13 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Flatulence: Change at follow-up (n=48, 46) | -0.7 (35.41) | 2.2 (34.00)
  Cachexia: Baseline (n=251, 253) | 33.1 (27.62) | 33.6 (26.84)
  Cachexia: Change at C2 D1 (n=197, 205) | 4.2 (24.26) | 0.6 (21.63)
  Cachexia: Change at C3 D1 (n=145, 157) | 4.6 (25.87) | -3.3 (21.13)
  Cachexia: Change at C4 D1 (n=101, 112) | 1.2 (26.37) | -6.2 (24.82)
  Cachexia: Change at C5 D1 (n=70, 64) | 0.5 (28.37) | -8.3 (24.48)
  Cachexia: Change at C6 D1 (n=40, 44) | -2.1 (24.80) | -5.3 (24.84)
  Cachexia: Change at C7 D1 (n=24, 26) | -0.7 (24.31) | -5.1 (25.27)
  Cachexia: Change at C8 D1 (n=10, 14) | 15.0 (34.64) | -4.7 (21.12)
  Cachexia: Change at C9 D1 (n=5, 6) | 16.7 (31.16) | 2.8 (19.47)
  Cachexia: Change at C10 D1 (n=1, 3) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (28.87)
  Cachexia: Change at C11 D1 (n=0, 1) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | -16.6 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Cachexia: Change at C12 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Cachexia: Change at C13 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Cachexia: Change at follow-up (n=48, 47) | 8.0 (31.69) | 6.4 (30.79)
  Side Effects: Baseline (n=209, 226) | 24.9 (21.21) | 27.4 (23.08)
  Side Effects: Change at C2 D1 (n=159, 181) | 11.2 (23.11) | 5.8 (22.06)
  Side Effects: Change at C3 D1 (n=113, 137) | 13.0 (24.67) | 4.7 (22.18)
  Side Effects: Change at C4 D1 (n=80, 102) | 10.1 (20.64) | 4.9 (22.48)
  Side Effects: Change at C5 D1 (n=54, 59) | 7.4 (25.55) | 3.6 (23.84)
  Side Effects: Change at C6 D1 (n=29, 40) | 8.1 (26.72) | -1.4 (25.32)
  Side Effects: Change at C7 D1 (n=17, 22) | 15.0 (20.77) | -1.0 (19.38)
  Side Effects: Change at C8 D1 (n=8, 11) | 9.7 (19.19) | -3.0 (22.83)
  Side Effects: Change at C9 D1 (n=3, 6) | 14.8 (23.15) | -1.9 (27.60)
  Side Effects: Change at C10 D1 (n=0, 3) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | 0.0 (40.12)
  Side Effects: Change at C11 D1 (n=0, 1) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | -33.4 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Side Effects: Change at C12 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Side Effects: Change at C13 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Side Effects: Change at follow-up (n=42, 42) | 18.8 (24.37) | 13.2 (27.80)
  Fear of Future Health (FH): Baseline (n=252, 250)) | 59.3 (31.33) | 61.1 (33.07)
  Fear of FH: Change at C2 D1 (n=192, 201) | -3.5 (31.82) | -9.6 (28.80)
  Fear of FH: Change at C3 D1 (n=145, 155) | -0.9 (34.02) | -11.6 (30.07)
  Fear of FH: Change at C4 D1 (n=103, 113) | -4.5 (32.70) | -15.9 (30.90)
  Fear of FH: Change at C5 D1 (n=71, 64) | -0.5 (31.12) | -10.9 (29.74)
  Fear of FH: Change at C6 D1 (n=42, 44) | -4.8 (30.86) | -14.4 (32.47)
  Fear of FH: Change at C7 D1 (n=27, 25) | -6.2 (22.72) | -13.3 (33.34)
  Fear of FH: Change at C8 D1 (n=12, 12) | 2.8 (30.02) | 5.6 (27.84)
  Fear of FH: Change at C9 D1 (n=6, 6) | 16.7 (27.90) | 16.7 (34.96)
  Fear of FH: Change at C10 D1 (n=2, 3) | -16.7 (23.62) | 11.1 (50.96)
  Fear of FH: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Fear of FH: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Fear of FH: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Fear of FH:Change at follow-up (n=48, 45) | 5.6 (28.63) | -4.4 (38.67)
  Future Plan ability: Baseline (n=250, 249) | 34.3 (33.59) | 38.0 (34.40)
  Future Plan ability: Change at C2 D1 (n=192, 198) | 6.1 (38.19) | -0.3 (34.58)
  Future Plan ability:Change at C3 D1 (n=142, 153) | 3.5 (39.65) | 0.4 (36.68)
  Future Plan ability:Change at C4 D1 (n=101, 112) | 5.6 (36.55) | 0.3 (37.04)
  Future Plan ability:Change at C5 D1 (n=70, 62) | 0.9 (34.05) | -3.8 (39.17)
  Future Plan ability:Change at C6 D1 (n=42, 42) | 4.8 (34.99) | 0.8 (46.27)
  Future Plan ability: Change at C7 D1 (n=26, 24) | 2.6 (28.18) | -7.0 (36.76)
  Future Plan ability: Change at C8 D1 (n=11, 11) | 6.1 (32.74) | 3.0 (43.36)
  Future Plan ability: Change at C9 D1 (n=5, 6) | 0.0 (23.55) | 0.0 (55.78)
  Future Plan ability: Change at C10 D1 (n=1, 3) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -11.1 (69.43)
  Future Plan ability: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Future Plan ability: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Future Plan ability: Change at C13 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Future Plan ability: Change at followup (n=48, 45) | 21.5 (35.40) | 5.2 (38.25)

7. Secondary Outcome: Change From Baseline Brief Pain Inventory-short Form (BPI-sf) Score
Description: BPI-sf is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-sf are 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each question is answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure can be scored by item, with lower scores being indicative of less pain or pain interference.
Time Frame: Baseline, Day 1 (D1) of each cycle (C2-C13) up to 28 days after the last dose (follow-up) or early withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Units on a scale
  Worst Pain: Baseline (n=247, 250) | 3.8 (2.84) | 3.7 (2.96)
  Worst Pain: Change at C2 D1 (n=192, 200) | -0.7 (3.04) | -0.9 (2.84)
  Worst Pain: Change at C3 D1 (n=138, 151) | -1.5 (3.09) | -0.9 (2.83)
  Worst Pain: Change at C4 D1 (n=99, 113) | -1.0 (3.41) | -0.9 (3.09)
  Worst Pain: Change at C5 D1 (n=69, 64) | -1.1 (3.43) | -1.2 (3.08)
  Worst Pain: Change at C6 D1 (n=41, 43) | -0.9 (2.98) | -1.0 (3.17)
  Worst Pain: Change at C7 D1 (n=25, 26) | -0.8 (2.27) | -0.9 (3.50)
  Worst Pain: Change at C8 D1 (n=12, 13) | 0.8 (2.56) | -1.5 (3.20)
  Worst Pain: Change at C9 D1(n=6, 6) | -1.8 (1.94) | -1.3 (1.51)
  Worst Pain: Change at C10 D1 (n=2, 3) | -2.0 (2.83) | -0.3 (2.31)
  Worst Pain: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Worst Pain: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Worst Pain: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Worst Pain: Change at follow-up (n=47, 46) | 0.5 (3.08) | 0.0 (3.21)
  Pain in Last 24 Hours (hrs): Baseline (n=246, 248) | 1.8 (1.92) | 1.7 (1.93)
  Pain in Last 24 hrs: Change at C2 D1 (n=193, 197) | -0.2 (2.21) | -0.3 (1.92)
  Pain in Last 24 hrs: Change at C3 D1 (n=138, 150) | -0.6 (2.01) | -0.3 (1.88)
  Pain in Last 24 hrs: Change at C4 D1 (n=99, 112) | -0.3 (2.15) | -0.0 (1.96)
  Pain in Last 24 hrs: Change at C5 D1 (n=69, 63) | -0.3 (2.41) | -0.2 (2.04)
  Pain in Last 24 hrs: Change at C6 D1 (n=40, 43) | -0.2 (2.07) | -0.1 (1.64)
  Pain in Last 24 hrs: Change at C7 D1 (n=25, 26) | 0.4 (1.47) | -0.0 (2.46)
  Pain in Last 24 hrs: Change at C8 D1 (n=12, 13) | 1.3 (2.34) | -0.2 (1.41)
  Pain in Last 24 hrs: Change at C9 D1 (n=6, 6) | -0.3 (1.37) | 0.2 (1.60)
  Pain in Last 24 hrs: Change at C10 D1 (n=2, 3) | -1.5 (2.12) | 0.3 (0.58)
  Pain in Last 24 hrs: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain in Last 24 hrs: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pain in Last 24 hrs: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain in Last 24 hrs: Change at followup (n=48, 45) | 0.4 (2.70) | 0.8 (2.58)
  Pain on the Average: Baseline (n=246, 248) | 2.9 (2.16) | 2.8 (2.27)
  Pain on the Average: Change at C2 D1 (n=195, 198) | -0.5 (2.02) | -0.5 (2.29)
  Pain on the Average: Change at C3 D1 (n=140, 149) | -0.8 (2.48) | -0.5 (2.10)
  Pain on the Average: Change at C4 D1 (n=99, 113) | -0.7 (2.44) | -0.6 (2.03)
  Pain on the Average: Change at C5 D1 (n=69, 63) | -0.7 (2.48) | -0.6 (2.29)
  Pain on the Average: Change at C6 D1 (n=40, 43) | -0.5 (2.07) | -0.9 (2.12)
  Pain on the Average: Change at C7 D1 (n=25, 26) | -0.3 (1.46) | -0.5 (2.97)
  Pain on the Average: Change at C8 D1 (n=12, 13) | 1.0 (2.00) | -1.4 (1.94)
  Pain on the Average: Change at C9 D1 (n=6, 6) | -1.7 (1.51) | -1.7 (1.86)
  Pain on the Average: Change at C10 D1 (n=2, 3) | -2.0 (2.83) | -1.0 (2.65)
  Pain on the Average: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain on the Average: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pain on the Average: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain on the Average: Change at followup (n=48, 45) | 0.6 (2.70) | 0.4 (2.74)
  Pain Right Now: Baseline (n=248, 249) | 2.1 (2.13) | 2.1 (2.36)
  Pain Right Now: Change at C2 D1 (n=196, 200) | -0.4 (2.23) | -0.5 (2.37)
  Pain Right Now: Change at C3 D1 (n=140, 150) | -0.8 (2.31) | -0.6 (2.06)
  Pain Right Now: Change at C4 D1 (n=99, 113) | -0.6 (2.26) | -0.5 (2.45)
  Pain Right Now: Change at C5 D1 (n=68, 63) | -0.5 (2.76) | -0.3 (2.65)
  Pain Right Now: Change at C6 D1 (n=40, 43) | -0.5 (1.96) | -0.5 (2.14)
  Pain Right Now: Change at C7 D1 (n=25, 26) | 0.1 (1.66) | -0.2 (3.26)
  Pain Right Now: Change at C8 D1 (n=12, 13) | 1.1 (1.93) | -0.6 (1.56)
  Pain Right Now: Change at C9 D1 (n=6, 6) | -1.5 (1.76) | -0.3 (0.52)
  Pain Right Now: Change at C10 D1 (n=2, 3) | -2.0 (2.83) | 0.7 (1.15)
  Pain Right Now: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain Right Now: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Pain Right Now: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain Right Now: Change at follow-up (n=48, 46) | 0.4 (2.64) | -0.0 (2.67)
  Relief Pain Treatment (Tx): Baseline (n=226, 221) | 7.8 (12.09) | 6.9 (9.71)
  Relief Pain Tx: Change at C2 D1 (n=164, 165) | 0.6 (13.96) | 0.4 (11.48)
  Relief Pain Tx: Change at C3 D1 (n=122, 124) | -2.1 (13.10) | 0.1 (9.16)
  Relief Pain Tx: Change at C4 D1 (n=88, 92) | -1.7 (13.51) | -0.9 (17.56)
  Relief Pain Tx: Change at C5 D1 (n=59, 51) | -2.9 (16.35) | 1.8 (11.62)
  Relief Pain Tx: Change at C6 D1 (n=34, 33) | -1.6 (11.90) | 0.5 (4.28)
  Relief Pain Tx: Change at C7 D1 (n=21, 18) | 1.0 (2.78) | -3.2 (19.65)
  Relief Pain Tx: Change at C8 D1 (n=10, 8) | -5.0 (21.20) | -11.6 (28.16)
  Relief Pain Tx: Change at C9 D1 (n=5, 5) | -14.0 (28.99) | -16.6 (35.44)
  Relief Pain Tx: Change at C10 D1 (n=1, 2) | 6.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (1.41)
  Relief Pain Tx: Change at C11 D1 (n=0, 1) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Relief Pain Tx: Change at C12 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Relief Pain Tx: Change at C13 D1 (n=0, 0) | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Relief Pain Tx: Change at follow-up (n=43, 36) | 0.2 (3.82) | -0.4 (5.08)
  General Activity: Baseline (n=243, 243) | 3.2 (3.11) | 3.0 (3.01)
  General Activity: Change at C2 D1 (n=190, 193) | -0.6 (2.96) | -0.7 (2.55)
  General Activity: Change at C3 D1 (n=135, 143) | -1.1 (3.47) | -0.7 (2.61)
  General Activity: Change at C4 D1 (n=97, 109) | -0.4 (3.10) | -0.8 (2.53)
  General Activity: Change at C5 D1 (n=66, 62) | -0.8 (3.64) | -0.5 (2.51)
  General Activity: Change at C6 D1 (n=40, 41) | -0.6 (3.82) | -0.7 (2.62)
  General Activity: Change at C7 D1 (n=25, 25) | -0.5 (2.87) | -0.4 (2.84)
  General Activity: Change at C8 D1 (n=12, 12) | 0.1 (2.07) | -0.8 (2.70)
  General Activity: Change at C9 D1 (n=6, 6) | -2.2 (2.71) | 0.3 (3.72)
  General Activity: Change at C10 D1 (n=2, 3) | -2.5 (3.54) | 3.0 (5.29)
  General Activity: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  General Activity: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  General Activity: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  General Activity: Change at follow-up (n=47, 44) | 1.0 (4.32) | 0.0 (3.63)
  Mood: Baseline (n=243, 241) | 3.0 (2.92) | 2.8 (2.77)
  Mood: Change at C2 D1 (n=191, 191) | -0.6 (2.74) | -0.2 (2.46)
  Mood: Change at C3 D1 (n=135, 141) | -1.0 (3.39) | -0.5 (2.51)
  Mood: Change at C4 D1 (n=98, 106) | -0.3 (3.22) | -0.9 (2.81)
  Mood: Change at C5 D1 (n=66, 61) | -0.7 (3.66) | -0.9 (2.59)
  Mood: Change at C6 D1 (n=40, 41) | -0.6 (3.23) | -0.8 (2.93)
  Mood: Change at C7 D1 (n=25, 25) | 0.0 (2.54) | -0.2 (3.18)
  Mood: Change at C8 D1 (n=12, 12) | 0.6 (1.31) | -1.1 (3.12)
  Mood: Change at C9 D1 (n=6, 6) | -1.3 (1.97) | -0.8 (3.31)
  Mood: Change at C10 D1 (n=2, 3) | -1.0 (1.41) | 3.3 (1.53)
  Mood: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Mood: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Mood: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Mood: Change at follow-up (n=47, 44) | 0.9 (3.65) | 0.2 (3.62)
  Walking Ability: Baseline (n=242, 243) | 2.2 (2.78) | 2.3 (2.81)
  Walking Ability: Change at C2 D1 (n=189, 194) | 0.1 (2.84) | -0.1 (2.61)
  Walking Ability: Change at C3 D1 (n=133, 143) | -0.2 (3.41) | -0.3 (2.52)
  Walking Ability: Change at C4 D1 (n=97, 108) | 0.3 (3.32) | -0.4 (2.64)
  Walking Ability: Change at C5 D1 (n=66, 62) | 0.1 (3.49) | -0.3 (2.37)
  Walking Ability: Change at C6 D1 (n=41, 41) | 0.5 (2.86) | -0.2 (2.24)
  Walking Ability: Change at C7 D1 (n=25, 25) | 1.1 (2.67) | -0.1 (2.42)
  Walking Ability: Change at C8 D1 (n=12, 12) | 0.7 (2.46) | -1.3 (2.42)
  Walking Ability: Change at C9 D1 (n=6, 6) | -1.0 (3.52) | 0.2 (4.62)
  Walking Ability: Change at C10 D1 (n=2, 3) | -2.0 (2.83) | 1.3 (5.51)
  Walking Ability: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Walking Ability: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Walking Ability: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Walking Ability: Change at follow-up (n=47, 45) | 0.9 (4.13) | 0.7 (3.27)
  Normal Work: Baseline (n=240, 240) | 3.5 (3.34) | 3.2 (3.23)
  Normal Work: Change at C2 D1 (n=187, 191) | -0.4 (3.24) | -0.1 (3.16)
  Normal Work: Change at C3 D1 (n=133, 139) | -0.6 (3.33) | -0.4 (2.67)
  Normal Work: Change at C4 D1 (n=96, 107) | -0.2 (3.15) | -0.7 (2.90)
  Normal Work: Change at C5 D1 (n=65, 61) | -0.7 (3.86) | -0.6 (2.71)
  Normal Work: Change at C6 D1 (n=39, 41) | 0.2 (3.62) | -0.2 (3.12)
  Normal Work: Change at C7 D1 (n=25, 24) | 0.5 (2.76) | -0.4 (2.52)
  Normal Work: Change at C8 D1 (n=12, 12) | -0.3 (3.70) | -0.1 (3.37)
  Normal Work: Change at C9 D1 (n=6, 6) | -1.5 (3.51) | 3.5 (4.32)
  Normal Work: Change at C10 D1 (n=2, 3) | -0.5 (0.71) | 1.3 (3.51)
  Normal Work: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Normal Work: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Normal Work: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Normal Work: Change at follow-up (n=46, 43) | 1.0 (4.54) | 0.3 (3.90)
  Relations: Baseline (n=244, 242) | 2.3 (2.93) | 1.9 (2.44)
  Relations: Change at C2 D1 (n=190, 193) | -0.3 (2.82) | 0.0 (2.18)
  Relations: Change at C3 D1 (n=136, 142) | -0.4 (3.81) | -0.0 (2.16)
  Relations: Change at C4 D1 (n=98, 108) | -0.2 (3.36) | -0.1 (2.52)
  Relations: Change at C5 D1 (n=66, 62) | -0.6 (3.11) | -0.1 (2.27)
  Relations: Change at C6 D1 (n=40, 41) | -0.3 (4.01) | -0.1 (2.76)
  Relations: Change at C7 D1 (n=25, 25) | 0.8 (3.32) | -0.7 (2.44)
  Relations: Change at C8 D1 (n=12, 12) | 0.6 (2.61) | -0.9 (2.35)
  Relations: Change at C9 D1 (n=6, 6) | -1.2 (2.93) | 0.8 (4.88)
  Relations: Change at C10 D1 (n=2, 3) | 1.0 (1.41) | 2.7 (2.52)
  Relations: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Relations: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Relations: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Relations: Change at follow-up (n=47, 45) | 0.7 (3.94) | 0.8 (3.56)
  Sleep: Baseline (n=244, 242) | 3.3 (3.16) | 3.2 (3.17)
  Sleep: Change at C2 D1 (n=191, 193) | -1.1 (3.36) | -0.9 (2.73)
  Sleep: Change at C3 D1 (n=136, 142) | -1.6 (3.52) | -1.1 (2.89)
  Sleep: Change at C4 D1 (n=98, 107) | -1.2 (3.29) | -1.2 (3.02)
  Sleep: Change at C5 D1 (n=66, 62) | -1.3 (4.06) | -0.8 (3.37)
  Sleep: Change at C6 D1(n=39, 41) | -1.5 (3.22) | -0.8 (3.62)
  Sleep: Change at C7 D1 (n=25, 25) | -0.2 (3.61) | -0.6 (2.81)
  Sleep: Change at C8 D1 (n=12, 12) | 0.6 (2.71) | -1.2 (3.51)
  Sleep: Change at C9 D1 (n=6, 6) | -2.3 (3.20) | 0.3 (2.07)
  Sleep: Change at C10 D1 (n=2, 3) | 1.0 (1.41) | 0.7 (3.51)
  Sleep: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Sleep: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Sleep: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Sleep: Change at follow-up (n=47, 44) | 0.5 (3.65) | -0.3 (3.54)
  Enjoyment of Life: Baseline (n=242, 240) | 3.5 (3.34) | 3.4 (3.17)
  Enjoyment of Life: Change at C2 D1 (n=191, 191) | -0.6 (2.99) | -0.5 (2.89)
  Enjoyment of Life: Change at C3 D1 (n=134, 142) | -0.7 (3.64) | -0.7 (2.77)
  Enjoyment of Life: Change at C4 D1 (n=98, 107) | -0.6 (3.58) | -0.9 (2.70)
  Enjoyment of Life: Change at C5 D1 (n=66, 62) | -0.6 (4.03) | -0.8 (3.07)
  Enjoyment of Life: Change at C6 D1 (n=40, 41) | -0.4 (3.87) | -1.0 (3.17)
  Enjoyment of Life: Change at C7 D1 (n=25, 25) | 0.4 (3.53) | -0.9 (2.28)
  Enjoyment of Life: Change at C8 D1 (n=12, 12) | 0.8 (2.98) | -0.8 (2.53)
  Enjoyment of Life: Change at C9 D1 (n=6, 6) | -0.5 (5.01) | 0.2 (2.86)
  Enjoyment of Life: Change at C10 D1 (n=2, 3) | 0.5 (0.71) | 2.3 (5.51)
  Enjoyment of Life: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Enjoyment of Life: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Enjoyment of Life: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Enjoyment of Life: Change at follow-up (n=47, 43) | 0.2 (3.68) | -0.2 (3.99)
  Combined Pain Intensity(PI): Baseline (n=248, 251) | 2.7 (1.98) | 2.6 (2.12)
  Combined PI: Change at C2 D1 (n=196, 202) | -0.4 (1.97) | -0.5 (1.97)
  Combined PI: Change at C3 D1 (n=140, 151) | -0.9 (2.15) | -0.6 (1.88)
  Combined PI: Change at C4 D1 (n=99, 114) | -0.6 (2.19) | -0.5 (1.99)
  Combined PI: Change at C5 D1 (n=69, 64) | -0.6 (2.46) | -0.6 (2.19)
  Combined PI: Change at C6 D1 (n=41, 43) | -0.5 (1.92) | -0.6 (1.89)
  Combined PI: Change at C7 D1 (n=25, 27) | -0.1 (1.48) | -0.4 (2.78)
  Combined PI: Change at C8 D1 (n=12, 13) | 1.0 (2.01) | -0.9 (1.76)
  Combined PI: Change at C9 D1 (n=6, 6) | -1.3 (1.51) | -0.8 (1.11)
  Combined PI: Change at C10 D1 (n=2, 3) | -1.9 (2.69) | -0.1 (1.44)
  Combined PI: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.5 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Combined PI: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Combined PI: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Combined PI:Change follow-up (n=48, 47) | 0.5 (2.34) | 0.2 (2.56)
  Combined Pain Interference(Pf):Baseline(n=244,243) | 3.0 (2.64) | 2.8 (2.52)
  Combined Pf: Change at C2 D1 (n=191, 194) | -0.5 (2.44) | -0.4 (1.97)
  Combined Pf: Change at C3 D1 (n=136,143) | -0.8 (2.99) | -0.5 (2.01)
  Combined Pf: Change at C4 D1 (n=98,109) | -0.4 (2.62) | -0.7 (2.12)
  Combined Pf: Change at C5 D1 (n=66, 62) | -0.6 (3.18) | -0.6 (2.07)
  Combined Pf: Change at C6 D1 (n=41, 41) | -0.4 (2.92) | -0.6 (2.38)
  Combined Pf: Change at C7 D1 (n=25, 25) | 0.3 (2.32) | -0.5 (2.10)
  Combined Pf: Change at C8 D1 (n=12, 12) | 0.4 (1.84) | -0.9 (2.15)
  Combined Pf: Change at C9 D1 (n=6, 6) | -1.4 (2.69) | 0.7 (2.86)
  Combined Pf: Change at C10 D1 (n=2, 3) | -0.5 (0.71) | 2.1 (2.90)
  Combined Pf: Change at C11 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.9 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Combined Pf: Change at C12 D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Combined Pf: Change at C13 D1 (n=1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -2.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Combined Pf: Change at follow-up (n=47, 45) | 0.7 (3.55) | 0.3 (3.40)

8. Secondary Outcome: Change From Baseline in Euro QoL Questionnaire- 5 Dimension (EQ-5D) Health State Profile
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Day 1 (D1) of each cycle (C2-C13) up to 28 days after the last dose (follow-up) or early withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Units on a scale
  Baseline (n=289, 290) | 0.665 (0.2709) | 0.690 (0.2479)
  Change at C2 D1 (n=231, 240) | 0.050 (0.2699) | 0.020 (0.2033)
  Change at C3 D1 (n=171, 178) | 0.053 (0.2528) | 0.028 (0.2362)
  Change at C4 D1 (n=128, 131) | 0.010 (0.2730) | 0.050 (0.2209)
  Change at C5 D1 (n=94, 80) | 0.010 (0.2889) | 0.044 (0.2092)
  Change at C6 D1 (n=57, 57) | 0.001 (0.2489) | 0.058 (0.2294)
  Change at C7 D1 (n=37, 36) | 0.049 (0.1891) | 0.075 (0.1838)
  Change at C8 D1 (n=17, 20) | -0.021 (0.2366) | 0.071 (0.2188)
  Change at C9 D1 (n=9, 9) | 0.049 (0.1878) | 0.121 (0.3006)
  Change at C10 D1 (n=3, 4) | 0.181 (0.2206) | 0.208 (0.3034)
  Change at C11 D1 (n=1, 1) | 0.000 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.058 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C12 D1 (n=1, 0) | 0.000 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at C13 D1 (n=1, 1) | 0.000 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.470 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at follow-up (n=65, 73) | -0.148 (0.3637) | -0.080 (0.3243)

9. Secondary Outcome: Change From Baseline in Euro QoL Questionnaire- 5 Dimension (EQ-5D) VAS Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Day 1 (D1) of each cycle (C2-C13) up to 28 days after the last dose (follow-up) or early withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Number analyzed (Participants) | 314 | 316
Millimeter (mm)
  Baseline (n= 277, 281) | 60.6 (23.67) | 62.6 (23.09)
  Change at Cycle 2 Day 1 (n= 223, 226) | 1.0 (19.64) | -0.4 (20.42)
  Change at Cycle 3 Day 1 (n= 161, 171) | 2.6 (22.30) | 1.1 (20.25)
  Change at Cycle 4 Day 1 (n=122, 128) | 0.5 (22.38) | 3.2 (19.81)
  Change at Cycle 5 Day 1 (n= 90, 79) | -0.3 (22.83) | 1.9 (19.40)
  Change at Cycle 6 Day 1 (n= 56, 56) | 1.0 (24.63) | 3.7 (21.84)
  Change at Cycle 7 Day 1 (n= 36, 35) | 2.6 (25.82) | 4.1 (22.52)
  Change at Cycle 8 Day 1 (n= 16, 19) | 3.8 (23.21) | 9.6 (28.55)
  Change at Cycle 9 Day 1 (n= 9, 9) | 22.2 (24.93) | 7.7 (20.00)
  Change at Cycle 10 Day 1 (n= 3, 4) | 20.0 (26.46) | 6.3 (24.62)
  Change at Cycle 11 Day 1 (n= 1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 30.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 12 Day 1 (n= 1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 13 Day 1 (n= 1, 1) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 36.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at follow-up (n= 62, 68) | -6.3 (24.07) | -4.8 (22.79)

10. Secondary Outcome: Population Pharmacokinetic (PK) Analysis for Axitinib (AG-013736)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1 (pre-dose), Day 29, Day 57 and then every 8 weeks up to 23 months
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: ng/mL

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE, both distinctly presented. An event may be categorized as SAE in 1 subject, AE in another or one subject may have experienced both serious and nonserious event. A participant randomized for Axitinib+Gemcitabine, received Gemcitabine only and was shifted to Placebo+Gemcitabine group for safety evaluation.
Arm/Group | Axitinib + Gemcitabine | Placebo + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 108/304 | 102/309
Other Adverse Events (participants affected / at risk) | 276/304 | 276/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Gemcitabine (N=304) | Placebo + Gemcitabine (N=309)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 10
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 3
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 9 | 11
Asthenia (General disorders) | 8 | 2
Chest pain (General disorders) | 1 | 0
Complication of device insertion (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
Device dislocation (General disorders) | 0 | 1
Device occlusion (General disorders) | 2 | 2
Disease progression (General disorders) | 9 | 15
Drug interaction (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 0
General physical health deterioration (General disorders) | 2 | 3
Generalised oedema (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Obstruction (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 13 | 5
Acholia (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 7 | 3
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 3 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Gallbladder necrosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3
Jaundice (Hepatobiliary disorders) | 6 | 4
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 2
Contrast media allergy (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Peritoneal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 5
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 3
Liver function test abnormal (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Diabetic coma (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Psychomotor skills impaired (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 3
Ureteric perforation (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 2
Phlebitis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Gemcitabine (N=304) | Placebo + Gemcitabine (N=309)
Anaemia (Blood and lymphatic system disorders) | 25 | 51
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Eosinopenia (Blood and lymphatic system disorders) | 1 | 0
Erythroblastosis (Blood and lymphatic system disorders) | 0 | 1
Erythropenia (Blood and lymphatic system disorders) | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 23 | 13
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 7
Neutropenia (Blood and lymphatic system disorders) | 73 | 53
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 48 | 34
Thrombocytosis (Blood and lymphatic system disorders) | 4 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 4 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Splinter haemorrhages (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 5
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Congenital foot malformation (Congenital, familial and genetic disorders) | 1 | 0
Auricular perichondritis (Ear and labyrinth disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 5 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 5
Hyperthyroidism (Endocrine disorders) | 2 | 1
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 15 | 4
Thyroiditis (Endocrine disorders) | 1 | 0
Asthenopia (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 3 | 0
Dry eye (Eye disorders) | 1 | 1
Eye pruritus (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 2 | 2
Ocular discomfort (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 2
Scotoma (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 12 | 12
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 54 | 52
Abdominal pain lower (Gastrointestinal disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 24 | 24
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 5 | 9
Cheilitis (Gastrointestinal disorders) | 4 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 88 | 91
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 96 | 64
Dry mouth (Gastrointestinal disorders) | 14 | 14
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 14 | 22
Dysphagia (Gastrointestinal disorders) | 7 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 2 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Faeces pale (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 8 | 9
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 4
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingival ulceration (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 6 | 1
Glossitis (Gastrointestinal disorders) | 7 | 0
Glossodynia (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 5
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Lip dry (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 138 | 112
Odynophagia (Gastrointestinal disorders) | 2 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 4 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Reflux gastritis (Gastrointestinal disorders) | 1 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Regurgitation (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 3 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1
Steatorrhoea (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 52 | 12
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 91 | 95
Adhesion (General disorders) | 0 | 1
Asthenia (General disorders) | 38 | 38
Catheter site erythema (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 2
Catheter site pruritus (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 2
Chest pain (General disorders) | 10 | 6
Chills (General disorders) | 13 | 11
Device occlusion (General disorders) | 0 | 1
Early satiety (General disorders) | 1 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 125 | 113
Feeling cold (General disorders) | 1 | 1
Feeling hot (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 6 | 2
Generalised oedema (General disorders) | 0 | 1
Hernia pain (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 1
Influenza like illness (General disorders) | 9 | 9
Injection site extravasation (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 2
Malaise (General disorders) | 0 | 2
Mass (Gastrointestinal disorders) | 1 | 0
Mucosal dryness (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 34 | 13
Oedema (General disorders) | 6 | 5
Oedema peripheral (General disorders) | 22 | 46
Pain (General disorders) | 16 | 7
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 38 | 44
Thirst (General disorders) | 2 | 1
Thrombosis in device (General disorders) | 2 | 0
Ulcer (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 4 | 4
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 2
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 6 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 9
Jaundice (Hepatobiliary disorders) | 3 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Liver tenderness (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 2
Contrast media allergy (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Acariasis (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 3 | 1
Candidiasis (Infections and infestations) | 2 | 0
Catheter site infection (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 3 | 4
Cystitis (Infections and infestations) | 4 | 3
Device related infection (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 1
Furuncle (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 7
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 6 | 5
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 3 | 1
Oral infection (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Perichondritis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 6 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 0 | 2
Septic encephalopathy (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 0
Skin candida (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 3 | 0
Tooth infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 2
Urinary tract infection (Infections and infestations) | 9 | 11
Viral infection (Infections and infestations) | 1 | 0
Anal injury (Injury, poisoning and procedural complications) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Burn oesophageal (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Alanine aminotransferase (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 29 | 24
Ammonia increased (Investigations) | 1 | 0
Aspartate aminotransferase (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 24 | 21
Bacterial test positive (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 2 | 1
Blood alkaline phosphatase (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 15 | 11
Blood amylase increased (Investigations) | 2 | 0
Blood bilirubin (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 6 | 9
Blood creatinine increased (Investigations) | 1 | 5
Blood culture positive (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 3 | 6
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 3
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 3 | 0
Blood sodium decreased (Investigations) | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2 | 1
Blood thyroid stimulating hormone increased (Investigations) | 16 | 0
Blood urea increased (Investigations) | 2 | 0
Blood urine (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 3 | 3
Eastern cooperative oncology group performance status worsened (Investigations) | 0 | 1
Electrocardiogram QRS complex abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin (Investigations) | 0 | 3
Haemoglobin decreased (Investigations) | 18 | 26
International normalised ratio increased (Investigations) | 1 | 2
Liver function test abnormal (Investigations) | 4 | 1
Lymph node palpable (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 6 | 4
Mean cell volume abnormal (Investigations) | 1 | 0
Monocyte count decreased (Investigations) | 2 | 0
Monocyte count increased (Investigations) | 0 | 1
Monocyte percentage increased (Investigations) | 1 | 0
Neutrophil count (Investigations) | 5 | 0
Neutrophil count decreased (Investigations) | 31 | 38
Neutrophil percentage decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count (Investigations) | 4 | 1
Platelet count decreased (Investigations) | 43 | 40
Platelet count increased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 1 | 1
Protein urine (Investigations) | 1 | 2
Protein urine present (Investigations) | 1 | 0
Prothrombin time abnormal (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 2
Prothrombin time shortened (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0
Red cell distribution width increased (Investigations) | 1 | 0
Thyroxine free increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 1
Tri-iodothyronine free increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 44 | 29
Weight increased (Investigations) | 0 | 2
White blood cell count (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 20 | 16
Decreased appetite (Metabolism and nutrition disorders) | 115 | 87
Dehydration (Metabolism and nutrition disorders) | 5 | 12
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 3 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 7
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 11
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Ageusia (Nervous system disorders) | 0 | 2
Amnesia (Nervous system disorders) | 3 | 2
Anaesthesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Cranial nerve disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 10 | 17
Dysaesthesia (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 25 | 14
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 45 | 26
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 6 | 2
Lethargy (Nervous system disorders) | 8 | 12
Loss of consciousness (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 4 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 7
Polyneuropathy (Nervous system disorders) | 1 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 3 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 16 | 19
Aversion (Psychiatric disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 7 | 3
Decreased activity (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 14 | 10
Dysphoria (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 2 | 3
Hallucinations, mixed (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 25 | 18
Loss of libido (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Vomiting psychogenic (Psychiatric disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 5 | 1
Haematuria (Renal and urinary disorders) | 4 | 4
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 4 | 3
Polyuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 17 | 12
Pyuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 1 | 0
Scrotal ulcer (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 19
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 68 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 20
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 1
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 9
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 17
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 43 | 41
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 4
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 10 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1
Abdominal cavity drainage (Surgical and medical procedures) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 4 | 9
Flushing (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 5 | 1
Hypertension (Vascular disorders) | 84 | 26
Hypotension (Vascular disorders) | 9 | 14
Orthostatic hypotension (Vascular disorders) | 2 | 0
Pallor (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 2 | 5
Phlebitis superficial (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 2 | 3
Vein pain (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.